CLINICAL TRIAL: NCT05707806
Title: Development and Validation of Learning and Decision-Making Tasks
Status: Recruiting | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001156; 001156-DA
Record Dates: First submitted 2023-01-31; First posted 2023-02-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01-05

CONDITIONS: Normal Physiology
Keywords: Behavioral Tasks; fMRI; Incentive Pocessing; Decision Making; Natural History

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy controls: generally healthy volunteers
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Enables the use of custom pulse sequence

SUMMARY:
Background:

Substance use disorders (SUD) can be considered disorders in the way people process incentives, learn, and make decisions. To understand why some people develop SUD, researchers need to develop reliable tests that show how people think and learn. This natural history study seeks to develop a set of tasks that could then be used to test how people learn and make decisions.

Objective:

To develop and validate behavioral tasks that could be used in future studies.

Eligibility:

Healthy people aged 18-45 years from the Baltimore area. They must also be enrolled in the NIDA screening protocol.

Design:

Participants will perform different tasks. Most tasks require 1-4 study visits; some may require up to 12. Visits are 1-14 days apart. All visits will last about 1-7 hours.

Participants will perform tasks on a computer. As they work they may be given different stimuli:

Smells. Participants will sniff odors through a plastic tube or mask on their nose.

Flavors. Participants will wear a mouthpiece and small amounts of different flavored liquids will be placed in their mouth.

Pictures. Participants will look at different images.

Sounds. Participants will wear headphones and various sounds will be played for them.

Food. Participants may be asked to eat a meal before, during, or after a task. The researchers will provide the meal.

During each task, participants will wear sensors to monitor their heart rate, blood pressure, breathing, and other physical changes in their bodies.

Some participants will have a functional magnetic resonance imaging (fMRI) scan. They will lie on a table that slides into a cylinder. They will perform tasks on a computer screen during the fMRI.

DETAILED DESCRIPTION:
Study Description:

From a behavioral perspective, substance-use disorders (SUD) can be considered as disorders of incentive processing, learning, and decision-making. The Learning and Decision-Making Unit at NIDA IRP conducts Basic Experimental Studies involving Humans (BESH) to study the neurocomputational mechanisms underlying these functions, and their disruption in SUD. For this, behavioral tasks suitable for use both in and outside the functional magnetic resonance imaging (fMRI) scanner need to be developed and validated.

Objectives:

The primary objective of this protocol is to develop and validate behavioral tasks inside and outside the fMRI scanner, and to determine their practical feasibility for future studies.

Endpoints:

The primary endpoint is to determine if the developed tasks reliably and appropriately measure specific cognitive functions, and if they yield measurable and interpretable fMRI results in the associated brain systems.

ELIGIBILITY:
* INCLUSION CRITERIA:

There are two levels of inclusion and exclusion criteria; those applying to all participants and those applying to participants in the MRI phase only. Participants will be cleared for both the behavioral and MRI phases, if eligible, and will be invited to sign one or both consents depending on what tasks are active at the time of consent. If a person is not MRI compatible, they will only be offered enrollment into the behavioral phase of the study.

In order to be eligible to participate in this study, an individual must meet the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18-45 years old. Justification: Many neural processes change with age, and these changes could introduce unwanted variability in both behavioral and MRI signals.
* In good general health.
* Agreement to adhere to Lifestyle Considerations throughout study duration

In order to be eligible to participate in the MRI phase of this study, an individual must - in addition - also meet all of the following criteria:

-Right-handed.

EXCLUSION CRITERIA:

Individuals who meet any of the following criteria will be excluded from participation:

* History of neurological illnesses or neurosurgery including but not limited to cerebrovascular accident, Parkinson disease, Alzheimer disease, Huntington disease, CNS tumor, significant head trauma with sequelae, multiple sclerosis or other demyelinating diseases, epilepsy, movement disorders. The MAI will also retain discretion to exclude based on a history of a neurological illness or trauma that may compromise data integrity.
* History of current (past 12 months) major DSM-5 psychiatric disorder including major affective disorder, obsessive-compulsive disorder, schizophrenia, or PTSD.
* Pattern of alcohol and drug use in the past 12 months that is indicative of harmful use, loss of control over use, or physical dependence.
* Daily nicotine, alcohol, or drug use (excluding caffeine) for at least 4 continuous weeks in the past 12 months.
* Current use of psychoactive medications and medications that affect alertness and that cannot (in principle) be withheld the night before the study visit. Participants who can withhold these medications will either (1) withhold the medication during this time or (2) not withhold the medication and pass a clinical assessment for intoxication on the day of the study visit. Based on participant preferences and MAI/PI judgement, participants who fail the clinical assessment for intoxication will either be withdrawn or rescheduled and asked to withhold the medication.
* For tasks that involve gustatory or olfactory stimuli, food intake: History of anaphylaxis, e.g., due to severe asthma or food and non-food allergies (e.g., latex, detergents, soap, etc.). This will disqualify participants for tasks that involve chemosensory stimuli or food intake, but not from the study itself.
* Uncorrected impairments in visual acuity.
* Non-English speaking. Justification: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify, given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI procedures. The inability to effectively communicate MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants.
* Pregnancy.
* Any other condition that in the judgment of the investigators is incompatible with participation.

An individual who meets any of the following criteria will be excluded from participation in the MRI phase of this study:

-Unable to undergo MRI scanning due to certain metallic or magnetic devices or implants in the body, or claustrophobia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: local community sample: metropolitan Baltimore area
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
task performance | each study visit
  to determine if the developed tasks reliably and appropriately measure specific cognitive functions, and if they yield measurable and interpretable fMRI results in the associated brain systems.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Kahnt, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share raw data from the study as this is a study to develop and validate behavioral tasks, to determine if they can reliably and appropriately measure specific functions, and if they yield measurable and interpretable fMRI results in the associated brain systems.